CLINICAL TRIAL: NCT00461773
Title: Randomized Phase II Study of Preoperative Letrozole (Femara) in Combination With Avastin in Hormone Receptor Positive Breast Cancer
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of recrual
Sponsor: Yale University (Other)
Collaborators: Novartis (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0609001793
Record Dates: First submitted 2007-04-16; First posted 2007-04-18 (Estimated); Results first posted 2021-03-16 (Actual); Last update posted 2021-03-16 (Actual); Status verified 2021-02

CONDITIONS: Hormone-Sensitive Breast Cancer; Breast Cancer
Keywords: Neoadjuvant treatment
MeSH Terms: conditions — Breast Neoplasms | interventions — Letrozole; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- bevacizumab (Active Comparator): brief exposure bevacizumab
  Interventions: Drug: Bevacizumab
- bevacizumab and letrozole (Active Comparator): brief exposure bevacizumab and letrozole
  Interventions: Drug: Letrozole; Drug: Bevacizumab

INTERVENTIONS:
Drug: Letrozole — Letrozole 2.5 mg po qd
  Other Names: Femara
  Arms: bevacizumab and letrozole
Drug: Bevacizumab — bevacizumab 10 mg/kg IV
  Other Names: Avastin

SUMMARY:
The purpose of this study is to evaluate the objective response rate of a combination of letrozole (Femara) and bevacizumab (Avastin) given preoperatively to postmenopausal patients with hormone sensitive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed operable or potentially operable invasive breast adenocarcinoma that is clinically palpable and measurable
* Age ≥ 18 years
* Clinical Stage T2-4, N0-3, M0 (Stage II-III)
* Postmenopausal defined as Age ≥ 60 years and/or Age >45 years with amenorrhea 12 months with an intact uterus and/or History of bilateral oophorectomy and/or FSH and estradiol levels in postmenopausal range
* ECOG PS 0, 1
* Unifocal disease
* ER and/or PR positive
* Adequate hematological, renal, and hepatic functions Absolute neutrophil count ≥ 1,500/µL Platelet count ≥ 100,000/µL creatinine ≤ 1.5 mg/dL Serum total bilirubin ≤ 1.5 mg/dL Alkaline phosphatase ≤ 3X the ULN for the reference lab SGOT/SGPT ≤ 3X the ULN for the reference lab
* Patients or their legal representatives must be able to read, understand and provide informed consent to participate in the trial
* Use of effective means of contraception (men and women) in subjects of child-bearing potential

Exclusion Criteria:

* Prior history of and/or therapy for invasive breast cancer (includes chemotherapy, radiation, hormonal therapy including AIs, tamoxifen, raloxifene, fulvestrant or any other antiestrogen/SERM)
* Clinically significant cardiovascular disease, EF <50%
* Known CNS disease
* History of deep vein thrombosis or pulmonary embolism
* Proteinuria at screening as demonstrated by either Urine protein:creatinine (UPC) ratio ≥ 1.0 at screening OR Urine dipstick for proteinuria ≥ 2+ (patients discovered to have ≥2+ proteinuria on dipstick urinalysis at baseline should undergo a 24 hour urine collection and must demonstrate ≤ 1g of protein in 24 hours to be eligible).
* Presence of non-healing wound or fracture
* Current, recent (within 4 weeks of the first infusion of this study), or planned participation in an experimental drug study other than a Genentech-sponsored bevacizumab cancer study
* Inadequately controlled hypertension (defined as systolic blood pressure >150 and/or diastolic blood pressure > 100 mmHg on antihypertensive medications)
* Any prior history of hypertensive crisis or hypertensive encephalopathy
* New York Heart Association (NYHA) Grade II or greater congestive heart failure (see Appendix E)
* History of myocardial infarction or unstable angina within 12 months prior to study enrollment
* Any history of stroke or transient ischemic attack at any time
* Significant vascular disease (e.g., aortic aneurysm, aortic dissection)
* Symptomatic peripheral vascular disease
* Evidence of bleeding diathesis or coagulopathy
* Major surgical procedure, open biopsy, or significant traumatic injury within 28 days prior to Day 0
* Core biopsy or other minor surgical procedures such as fine needle aspirations or core biopsies within 7 days prior to Day 0
* Pregnant (positive pregnancy test) or lactating. Use of effective means of contraception (men and women) in subjects of child-bearing potential is mandatory
* History of abdominal fistula, gastrointestinal perforation, or intra-abdominal abscess within 6 months prior to Day 0
* Known hypersensitivity to any component of bevacizumab or letrozole
* Inability to comply with study and/or follow-up procedures

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2007-03; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gina Chung, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University, Yale Cancer Center, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Bevacizumab and Letrozole: brief exposure bevacizumab and letrozole
  Letrozole: Letrozole 2.5 mg once orally daily
  Bevacizumab: bevacizumab 10 mg/kg IV
Period: Overall Study
Arm/Group | Bevacizumab | Bevacizumab and Letrozole
Started | 3 | 2
Completed | 3 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bevacizumab | Bevacizumab and Letrozole | Total
Number analyzed (Participants) | 3 | 2 | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 2 | 4
  >=65 years | 1 | 0 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 2 | 5
  Male | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Patients With Objective Tumor Response
Description: Clinical objective tumor response with 14 weeks of Neoadjuvant Letrozole combined with Bevacizumab was assessed using the following categories:
  Complete Response (CR): tumor is no longer visible. Partial response (PR): ≥ 50% decrease from baseline in the product of two perpendicular diameters, no new lesions. Progressive disease (PD): ≥ 25% increase of the product of two perpendicular diameters or new lesions. Stable Disease (SD): Neither CR, PR, or PD criteria met. Clinical tumor assessment was performed at baseline and every 2 weeks until week 18 prior to definitive surgery.
Time Frame: Up to 18 weeks
Population: All patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab | Bevacizumab and Letrozole
Number analyzed (Participants) | 3 | 2
Participants
  Complete Response | 1 | 0
  Partial Response | 2 | 1
  Progressive Disease | 0 | 0
  Stable Disease | 0 | 1

2. Secondary Outcome: Breast Conservation
Description: To assess breast conservation (actual surgery performed and baseline feasible surgery) of 14 weeks of neoadjuvant letrozole combined with bevacizumab.
  At baseline and immediately prior to surgery, the investigator will record the extent of the least invasive feasible surgery option at that time point, according to the following categories: 1. Breast conserving surgery is feasible; 2. A mastectomy is needed; 3. Tumor is inoperable, but potentially operable after neoadjuvant treatment.
  Following surgery, the investigator will record the extent of the actual surgery performed according to the following categories:
  1. Breast conserving surgery performed; 2. Mastectomy performed 3. No surgery performed (reason should be specified).
Time Frame: Up to 14 weeks
Population: All patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab | Bevacizumab and Letrozole
Number analyzed (Participants) | 3 | 2
Participants
  Breast Conservation Feasible Baseline: number analyzed (Participants) | 2 | 1
  Breast Conservation Feasible Baseline: Performed at 14 weeks | 2 | 1
  Breast Conservation Feasible Baseline: Not Performed at 14 weeks | 0 | 0
  Mastectomy Needed at Baseline: number analyzed (Participants) | 1 | 1
  Mastectomy Needed at Baseline: Performed at 14 weeks | 1 | 1
  Mastectomy Needed at Baseline: Not Performed at 14 weeks | 0 | 0

3. Secondary Outcome: Radiographic Tumor Response
Description: To assess radiographic tumor response after 14 weeks of Neoadjuvant Letrozole combined with Bevacizumab, mammogram were performed at baseline and at week 18 prior to definitive surgery.
  Tumors response was assessed using RECIST criteria RECIST:
  CR: Tumor is no longer visible PR: ≥ 30% decrease from baseline in the longest diameter, no new lesions PD: ≥ 20% increase in longest diameter recorded or new lesions SD: Neither CR, PR, or PD criteria met
Time Frame: 18 weeks
Population: All patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab | Bevacizumab and Letrozole
Number analyzed (Participants) | 3 | 2
Participants
  CR | 0 | 0
  PR | 2 | 2
  PD | 0 | 0
  SD | 1 | 0

4. Secondary Outcome: Pathologic Complete Response
Description: To assess pathologic complete response after 14 Weeks of Neoadjuvant Letrozole combined with Bevacizumab, the pathologic response was determined on the surgically excised specimen at the time of definitive surgery.
  The size of the residual tumor would be measured grossly if possible and confirmed microscopically.
  The excised residual tumor was be assessed using RECIST criteria.
  RECIST:
  CR: Tumor is no longer visible PR: ≥ 30% decrease from baseline in the longest diameter, no new lesions PD: ≥ 20% increase in longest diameter recorded or new lesions SD: Neither CR, PR, or PD criteria met
Time Frame: Up to 18 weeks
Population: All patients.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab | Bevacizumab and Letrozole
Number analyzed (Participants) | 3 | 2
Participants
  CR | 0 | 0
  PR | 1 | 1
  PD | 1 | 1
  SD | 1 | 0

5. Secondary Outcome: Tumor Response With Biological Correlates
Description: To correlate response with biological correlates detected at baseline and after 1 cycle of treatment with either Bevacizumab alone or Bevacizumab combined with Letrozole.
Time Frame: 2 weeks
Population: These labs were never conducted as the study was terminated after 5 patients.
Arm/Group | Bevacizumab | Bevacizumab and Letrozole
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Drug Tolerability
Description: To assess the tolerability of 14 weeks of Neoadjuvant Letrozole combined with Bevacizumab, individual toxicities were graded according to the National Cancer Institute (NCI) Common Toxicity Criteria (CTC) Version 3.0. Information about all adverse events, whether volunteered by the subject, discovered by investigator questioning, or detected through physical examination, laboratory test or other means, were collected and recorded on the Adverse Event Case Report Form and followed as appropriate. An adverse event (AE) is any undesirable sign, symptom or medical condition occurring after starting study drug (or therapy) even if the event is not considered to be related to study drug (or therapy). Study drug (or therapy) includes the drug (or therapy) under evaluation, and any reference or placebo drug (or therapy) given during any phase of the trial. AE's graded 3 or 4 would be considered serious and be reported as measures of tolerability.
Time Frame: Up to 18 weeks
Population: All adverse events are presented in the adverse event module.
Measure: Count of Participants; unit: Participants
Arm/Group | Bevacizumab | Bevacizumab and Letrozole
Number analyzed (Participants) | 3 | 2
Participants
  Any Grade 3 Adverse Events | 0 | 0
  Any Grade 4 Adverse Events | 0 | 0

ADVERSE EVENTS:
Time Frame: Up to 18 weeks
Arm/Group | Bevacizumab | Bevacizumab and Letrozole
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/2
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/2
Other Adverse Events (participants affected / at risk) | 3/3 | 2/2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bevacizumab (N=3) | Bevacizumab and Letrozole (N=2)
ALLERGY/IMMUNOLOGY (Immune system disorders) | 2 (4) | 0 (0)
AUDITORY/EAR (Ear and labyrinth disorders) | 0 (0) | 1 (1)
BLOOD/BONE MARROW (Blood and lymphatic system disorders) | 0 (0) | 1 (3)
CARDIAC GENERAL (Cardiac disorders) | 2 (2) | 2 (4)
CONSTITUTIONAL SYMPTOMS (General disorders) | 2 (10) | 2 (8)
DERMATOLOGY/SKIN (Skin and subcutaneous tissue disorders) | 2 (9) | 2 (3)
ENDOCRINE (Endocrine disorders) | 1 (1) | 1 (4)
GASTROINTESTINAL (Gastrointestinal disorders) | 2 (9) | 2 (8)
HEMORRHAGE/BLEEDING (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
LYMPHATICS (Immune system disorders) | 1 (1) | 0 (0)
METABOLIC/LABORATORY (Metabolism and nutrition disorders) | 3 (29) | 2 (20)
MUSCULOSKELETAL/SOFT TISSUE (Musculoskeletal and connective tissue disorders) | 1 (2) | 1 (1)
NEUROLOGY (Nervous system disorders) | 1 (1) | 1 (9)
OCULAR/VISUAL (Eye disorders) | 1 (1) | 2 (2)
PAIN (General disorders) | 3 (17) | 2 (16)
PULMONARY/UPPER RESPIRATORY (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 2 (5)
RENAL/GENITOURINARY (Renal and urinary disorders) | 1 (1) | 0 (0)
SYNDROMES (General disorders) | 1 (1) | 0 (0)
VASCULAR (Vascular disorders) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The data reported are summaries of the available data that were collected up until the time of study termination.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes